CLINICAL TRIAL: NCT03171090
Title: Efficacy of Bilaterally Ultrasonic Guided Sphenopalatine Ganglion Block for Perioperative Pain Management in Maxilofacial Cancer Surgeries
Brief Title: Efficacy of Bilateral Ultrasonic Guided Sphenopalatine Ganglion Block in Maxilofacial Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed H Othman, Associte professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IORG0003381
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Maxillofacial Tumors
MeSH Terms: interventions — Anesthetics, Local; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sphenopalatine block using local anasthetic (Active Comparator)
  Interventions: Other: sphenopalatine block with saline
- sphenopalatine block using saline (Placebo Comparator)
  Interventions: Other: sphenopalatine block with local anesthetic

INTERVENTIONS:
Other: sphenopalatine block with local anesthetic — bilateral ultrasonic guided sphenopalatine ganglion block using local anesthetic after induction of general anesthesia in maxilofacial cancer surgeries
  Arms: sphenopalatine block using saline
Other: sphenopalatine block with saline — bilateral ultrasonic guided sphenopalatine ganglion block using saline after induction of general anesthesia in maxilofacial cancer surgeries
  Arms: sphenopalatine block using local anasthetic

SUMMARY:
Patients will be randomly allocated according to computer - generated tables to one of two groups, group (A) ultrasonic guided sphenopalatine block using local anasthetic, group (B) ultrasonic guided sphenopalatine block using saline. Before induction anesthesia the following will be assessed, time needed to perform the technique, time till onset of the block, distribution of the block (Opthalmic, Maxillary, Mandibular) by needle brick.Intra and post- operatively the following will be assesse the quality of operative filed every 30 min intra-operatively using a pre- defined average category scale (ACS) (from 0 to 5), End tidal Sevo Flurane concentration will be recorded intra- operatively every 5 minutes, The total amount of Nitroglycerine used to achieve the target MAP and frequency of propranolol usage will be recorded,emergence time, postoperative VAS score and amount of meperdine used for rescue analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients of ASA physical status I and II, aged 20-70 year who will be scaduled for Maxillo - facial cancer surgeries

Exclusion Criteria:

* patients with disfigurement and disturbed anatomy that will not allow easy access to the sphenopalatine ganglion, bleeding disorders, history of hepatic, renal or cardiopulmonary dysfunction, patients receiving drugs affecting coagulation or cardiovascular active medication are excluded also patients having infection or allergies to local anesthetics

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Post - operative analgesia | 24 hours postopeatively
  according to VAS measured in the postoperative period

SECONDARY OUTCOMES:
total dose of analgesic consumption | 24 hours
  total nalufen dose
number of patients required analgesia | 24 hours
  number of patients required nalufen

CONTACTS AND LOCATIONS:
Locations (1):
- NCI, Cairo university, Cairo, Egypt